CLINICAL TRIAL: NCT00224757
Title: Transesophageal Echocardiography to Identify pAtients With Low Risk of Stroke in Atrial Fibrillation
Brief Title: Transesophageal Echocardiography to Identify pAtients With Low Risk of Stroke in Atrial Fibrillation - TIARA Pilot Study
Acronym: TIARA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Interuniversity Cardiology Institute of the Netherlands (Other Government)
Responsible Party: Principal Investigator, NHT Dinh, Drs., The Interuniversity Cardiology Institute of the Netherlands
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0415
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: Echocardiography
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin (Active Comparator): Ascal 100mg once daily
  Interventions: Procedure: Transoesophageal echocardiography
- Coumarin derivates (Active Comparator): Acenocoumarol or fenprocoumon
  Interventions: Procedure: Transoesophageal echocardiography

INTERVENTIONS:
Procedure: Transoesophageal echocardiography — TEE
  Other Names: No other names

SUMMARY:
In this multi centre pilot study we will perform TEE in patients with AF who are eligible for VKA treatment. TTE will be used as pre-screening: if TTE shows left atrial abnormalities or aortic plaque, patients will be excluded from randomisation. TEE will be performed in all other patients to detect or exclude complex aorta plaques or signs of left atrial stasis. Three hundred patients who do not have these features on TTE will be randomly assigned to treatment with aspirin or VKA. Follow-up will be 1 year.

DETAILED DESCRIPTION:
BACKGROUND Atrial fibrillation (AF) is an independent risk factor for stroke. Therapy with vitamin K antagonists (VKA) and aspirin reduces the risk of thromboembolism (TE) dramatically. Risk stratification is nowadays based on clinical characteristics. However, many high risk AF patients may actually be at low risk, identified by trans-oesophageal echocardiography (TEE).

HYPOTHESIS A comprehensive strategy of TEE based aspirin treatment in AF patients eligible for VKA therapy is safe and feasible.

OBJECTIVES

1. To show that TEE based aspirin treatment is safe when compared with VKA therapy.
2. To test the feasibility of TEE as a tool to detect all four echocardiographic features of high stroke risk.

METHODS In this multi centre pilot study we will perform TEE in patients with AF who are eligible for VKA treatment. TTE will be used as pre-screening: if TTE shows left atrial abnormalities or aortic plaque, patients will be excluded from randomisation. TEE will be performed in all other patients to detect or exclude complex aorta plaques or signs of left atrial stasis. Three hundred patients who do not have these features on TTE will be randomly assigned to treatment with aspirin or VKA. Follow-up will be 1 year.

EXPECTED RESULTS Application of a new echo-guided antithrombotic strategy as proposed herein is feasible and may help to reduce bleeding whilst stroke prevention is maintained. If the lower limit of the 95% confidence interval of the yearly incidence of the primary endpoint on aspirin remains below 4.4% then a large multi centre randomised controlled trial will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Documented atrial fibrillation or atrial flutter, paroxysmal or permanent
* Conventional indication for VKA treatment
* Signed informed consent

Exclusion Criteria:

* Planned electro cardioversion
* Very high risk of TE (previous ischemic stroke or systemic TE, symptoms of heart failure or left ventricular dysfunction, mitral valve stenosis, hypertrophic cardiomyopathy)
* Indication for VKA treatment other than atrial fibrillation (e.g. mechanic valve prosthesis)
* Atrial fibrillation secondary to reversible diseases (e.g. thyrotoxicosis)
* Contraindication for treatment with VKA, aspirin, or clopidogrel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2005-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
A composite of the following endpoints: ischemic stroke, systemic embolism, major bleeding, acute coronary syndrome, death. | at least 1 year

SECONDARY OUTCOMES:
Completion of a technical adequate TTE/TEE on the four echocardiographic features of high stroke risk. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: HJGM Crijns, MD, PhD, Study Chair — Academisch Ziekenhuis Maastricht
Locations (10):
- Netherlands (10):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Twenteborg, Almelo
  - VUMC, Amsterdam
  - Rijnstate Ziekenhuis, Arnhem
  - Amphia Ziekenhuis, Breda
  - Atrium Medisch Centrum Heerlen, Heerlen
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Diaconessenhuis Meppel, Meppel
  - UMCN, Nijmegen
  - Viecuri, Venlo